CLINICAL TRIAL: NCT04251130
Title: Linking Tau PET to Medial Temporal Lobe Subregions With High Resolution MRI
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 833864
Record Dates: First submitted 2020-01-03; First posted 2020-01-31 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — ((18)F)PI-2620

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cognitively Normal Older Adults: Subjects will receive an IV bolus injection of approximately 5 mCi ± 20% of [18F]PI-2620. All subjects will undergo a 30-minute brain PET/CT scan performed starting at approximately 45 minutes' post injection of [18F]PI-2620. A low-dose CT scan will be acquired according to standard PET/CT imaging procedures to be used for attenuation correction. All images will be reconstructed using standard reconstruction techniques
  Interventions: Drug: 2-(2-([18F]fluoro)pyridin-4-yl)-9H-pyrrolo[2,3-b:4,5-c']dipyridine
- Mild Cognitively Impaired Older Adults or Older Adults with Alzheimer's Disease: Subjects will receive an IV bolus injection of approximately 5 mCi ± 20% of [18F]PI-2620. All subjects will undergo a 30-minute brain PET/CT scan performed starting at approximately 45 minutes' post injection of [18F]PI-2620. A low-dose CT scan will be acquired according to standard PET/CT imaging procedures to be used for attenuation correction. All images will be reconstructed using standard reconstruction techniques
  Interventions: Drug: 2-(2-([18F]fluoro)pyridin-4-yl)-9H-pyrrolo[2,3-b:4,5-c']dipyridine

INTERVENTIONS:
Drug: 2-(2-([18F]fluoro)pyridin-4-yl)-9H-pyrrolo[2,3-b:4,5-c']dipyridine — A small molecule aimed for binding and PET-imaging of aggregated tau protein in the human brain.
  Other Names: [18F]PI-2620

SUMMARY:
The investigators will conduct a tau PET scan in cognitively normal older adults and patients with Mild Cognitive Impairment (MCI), enrolled in the National Alzheimer's Coordinating Center (NACC) study at the University of Pennsylvania's Penn Memory Center/Alzheimer's Disease Core Center (PMC/ADC).

DETAILED DESCRIPTION:
This is a cross-sectional and longitudinal study using the radiotracer [18F]-PI-2620 to determine the relationship of tau pathology to both cross-sectional and longitudinal clinical and biomarker data of NACC cohort participants who are Cognitively Normal or MCI. All subjects will already be part of the longitudinal cohort study, known as the "NACC" cohort, of the PMC/ADC (protocol 068200). Participants will provide informed consent for this protocol before beginning any study procedures. After screening assessments, participants will undergo PET scan imaging with [18F]PI-2620. There will be one follow-up [18F]PI-2620 PET scan approximately 18 +/- 6 months after bas eline scan.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 60 years of age.
* Part of the NACC longitudinal cohort (IRB# 068200) of the PMC/ADCC with consensus conference designation of cognitively normal or Mild Cognitive Impairment (MCI) or Alzheimer's Disease (AD) Possible or Probable.
* NACC longitudinal visit completed or scheduled within 6 months before or after enrollment in this study.
* Women must be post-menopausal or surgically sterile.
* An amyloid PET scan, completed as a part of the NACC protocol (IRB# 825943), must be performed or scheduled within 12 months before or after the [18F]PI-2620 PET scan.
* A brain MRI, completed as a part of NACC protocol (IRB# 068200), must be performed or scheduled within 6 months before or after the [18F]PI-2620 PET scan. Scan should be of adequate research quality, including 3 Tesla and/or 7 Tesla high-resolution imaging of MTL structure.

Exclusion Criteria:

* Have any medical or psychiatric conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.
* Have evidence of structural abnormalities such as major stroke or mass on MRI that is likely to interfere with analysis of the PET scan.
* Inability to tolerate or contraindication to imaging procedures in the opinion of an investigator or treating physician.
* Have a history of significant or ongoing alcohol abuse or substance abuse or dependence based on medical record review or self-reported.

The inclusion / exclusion criteria will be ascertained through self-report in conjunction with any medical history available through the participant's medical or research records (EPIC or the ADC database)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults cognitively normal or Mild Cognitive Impairment (MCI) or Alzheimer's Disease.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-03-11 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between PI-2620 SUVR and MTL subregion thickness | Baseline
  Correlation between cross-sectional PI-2620 standard uptake value ratio (SUVR) and MTL subregion thickness (mm) in both controls and MCI/AD.
Interaction between PI-2620 SUVR and amyloid status prediction of MTL subregion thickness | Baseline
  Interaction between cross-sectional PI-2620 standard uptake value ratio (SUVR) and amyloid status for prediction of MTL subregion thickness (mm) in both controls and MCI/AD.
Correlation between longitudinal PI-2620 SUVR and MTL subregion thickness | 18-24 months
  Correlation between longitudinal PI-2620 standard uptake value ratio (SUVR) and MTL subregion thickness (mm) in both controls and MCI/AD.
Interaction between longitudinal PI-2620 SUVR and amyloid status for prediction of MTL subregion thickness | 18-24 months
  Interaction between longitudinal PI-2620 standard uptake value ratio (SUVR) and amyloid status for prediction of MTL subregion thickness (% annual change) in both controls and MCI/AD.

CONTACTS AND LOCATIONS:
Overall Officials: David Wolk, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, School of Medicine, Philadelphia, Pennsylvania, United States